CLINICAL TRIAL: NCT06741462
Title: Prospective Randomized Study to Prove a Positive Care Effect of the Digital Health Assistant ADELE A0004 for Patients with a Care Level
Brief Title: Positive Care Effect of the Digital Health Assistant ADELE for Patients with Care Level
Acronym: A0004
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Phil Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APH01_PG
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Care Givers; Health; Care of the Elderly; Health Care Delivery; Mobility and Independence
Keywords: digital health; health assistant; Patient autonomy; care level

STUDY DESIGN:
Intervention Model Description: Intervention group: Participants in the intervention group were patients with proven care level who had been provided ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were gathered using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1). Control group: Participants in the control group were patients with proven care level who were not provided with ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were collected using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1).
  In addition, after the end of the observation period (from t0 to t1), the participants in the control group were offered an extension of a further 3 months on average using ADELE (from t1 to t2).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Participants in the intervention group were patients with proven care level who had been provided ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were gathered using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1).
  Interventions: Device: Digital health assistant ADELE A0004
- Control Group (No Intervention): Participants in the control group were patients with proven care level who were not provided with ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were collected using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1). In addition, after the end of the observation period (from t0 to t1), the participants in the control group were offered an extension of a further 3 months on average using ADELE (from t1 to t2).

INTERVENTIONS:
Device: Digital health assistant ADELE A0004 — The digital health assistant ADELE A0004 (ADELE for short) improves the daily lives of patients with care level and enables them to deal better and more independently with the everyday burdens resulting from the need for care. Participants in the intervention group were provided with ADELE to use during the study period for e.g., tracking of daily reminders, voice-based recording, interpretation and classification of their vital signs and body conditions.
  Arms: Intervention Group

SUMMARY:
Care is becoming an increasingly important topic in Germany due to the rising number of people in need of care. There are currently around 5 million people with a care level in Germany who are permanently dependent on help to cope with everyday life due to health impairments. The risk of needing care increases with age. ALMA PHIL has set itself the goal of using the digital health assistant ADELE A0004 (ADELE for short) to make everyday life easier for people in need of care, thereby maintaining their independence and preventing any deterioration in their need for care.

The study aims to prove the positive care benefits of using ADELE for people with a care level on e.g., the improvement and stabilization of independence especially in the home care situation; reducing the mental and physical strain of coping with the need for care in everyday life; improving the mobility of the person in need of care; maintaining cognitive and communicative abilities and on the improvement of adherence. In addition, the nursing benefits of ADELE also include relieving the daily burden on the personal care network.

DETAILED DESCRIPTION:
Care is becoming an increasingly important topic in Germany due to the rising number of people in need of care. There are currently around 5 million people with a care level in Germany who are permanently dependent on help to cope with everyday life due to health impairments. The risk of needing care increases with age. While around 9% of people aged 70 to 74 living in Germany are in need of care, the proportion for those aged 90 and over is around 82%. The forecasts of the Federal Statistical Office also show a growing number of people with a care level in the coming years and an associated increase in the need for care. Around four out of five people in need of care are nursed at home, mostly by relatives.

ALMA PHIL has set itself the goal of using the digital health assistant ADELE A0004 (ADELE for short) to make everyday life easier for people in need of care, thereby maintaining their independence and preventing any deterioration in their need for care.

This study aims to prove the positive care benefits of using ADELE for people with a care level. The increase in knowledge from the study consists in the positive effectiveness and the nursing benefits for people in need of care, e.g., on the improvement and stabilization of independence especially in the home care situation; on reducing the mental and physical strain of coping with the need for care in everyday life; on improving the mobility of the person in need of care; on maintaining cognitive and communicative abilities (independence and social interaction) and on the improvement of adherence (regular intake of medication, regular fulfillment of set goals). In addition, the nursing benefits of ADELE also include relieving the daily burden on the personal care network.

A prospective randomized multicenter study with a parallel group design was used. To conduct the study, adult participants with proven care level were randomly assigned to the intervention group or the control group as part of a 1:1 randomization. The observation period per participant was 3 months on average. The data was collected by means of questionnaires. ADELE was provided to the intervention group. ADELE was not provided to the participants in the control group.

The primary objective of the study was to prove the improvement in patient sovereignty from the perspective of the patient with a care level, measured after 3 months. As secondary endpoints were defined (all measured after 3 months): the improvement of mobility, the improvement of mental and physical health, the improvement in patient sovereignty from the perspective of the caregiver, the reducing of the burden on the caregiver of the person in need of care in everyday life through the digital care application. As additional exploratory endpoints were the improvement in health confidence and the reduction of the systolic and diastolic blood pressure values defined, measured after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Age (at least 18 years)
* Level of care I-V: People in need of care with impaired cognitive abilities; People in need of care with impaired ability to structure their day and/or impaired ability to remember; People in need of care with impaired ability to orient themselves in time; Risk of falls in the normal everyday environment
* Person must be able to understand the patient information
* Written declaration of consent is signed at the beginning of interview 1

Exclusion Criteria:

* Age under 18 years
* Persons belonging to specially protected groups (e.g. persons temporarily or permanently unable to give consent)
* Person suffers from mental illness that prevents them from understanding the information about the study, giving their consent or complying with the requirements of the study
* Person is unable to operate the application properly
* Person has already had contact with the application and/or a comparable application
* Person is participating in another study
* Emergency and intensive care medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Change of patient autonomy | From enrollment to the end of treatment at 3 months
  Change of patient autonomy, defined as the stabilization of autonomous coping with burdens in everyday life from the perspective of the patient with a care level, measured after 3 months based on PS19 score. The PS19 questionnaire had 19 items. The score is between 0 (Minimum) and 57 (Maximum). A higher value is better.

SECONDARY OUTCOMES:
Change in mobility of patient | From enrollment to the end of treatment at 3 months
  Evaluation of the 6-minute walk test (short 6MWT) to assess the performance of the patient with a care level and to be able to monitor it over time. A higher value is better.
Change of patient autonomy | From enrollment to the end of treatment at 3 months
  Change of patient autonomy, defined as the stabilization of autonomous coping with burdens in everyday life from the perspective of the patient with a care level, measured after 3 months based on PS8D score. The PS8D questionnaire had 8 items. The score is between 0 (Minimum) and 24 (Maximum). A higher value is better.
Change of patient autonomy (caregiver perpective) | From enrollment to the end of treatment at 3 months
  Change of autonomy of patient with care level, defined as the stabilization of autonomous coping with burdens in everyday life from the perspective of the caregiver, measured after 3 months based on PS8D-P score. The PS8D-P questionnaire had 8 items. The score is between 0 (Minimum) and 24 (Maximum). A higher value is better.
Change of patient autonomy (caregiver perpective) | From enrollment to the end of treatment at 3 months
  Change of autonomy of patient with care level, defined as the stabilization of autonomous coping with burdens in everyday life from the perspective of the caregiver, measured after 3 months based on PS19-P score. The PS19-P questionnaire had 19 items. The score is between 0 (Minimum) and 57 (Maximum). A higher value is better.
Change of Reliefe for caregiver | From enrollment to the end of treatment at 3 months
  Relieving the caregiver of the person in need of care in everyday life through the digital care application, measured after 3 months based on the ICG score. The ICG questionnaire had 6 items. The score is between 0 (Minimum) and 18 (Maximum). A higher value is better.
Change of health condition | From enrollment to the end of treatment at 3 months
  Change of health condition, measured after 3 months using Short Form 12 Health Survey (SF-12). The scale is based on 12 items. The score is between 0 (Minimum) and 100 (Maximum). A higher value is better.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoffmann, Prof. Dr. med., Study Chair — (Minority) shareholder; Oliver Vonend, Prof. Dr. med., Principal Investigator; Hans-Peter Reiffen, Prof. Dr. med., Study Director
Locations (2):
- Germany (2):
  - Ökumenische Sozialstation Heidenheimer Land, Heidenheim, Baden-Wurttemberg
  - Johanniter-Unfall-Hilfe e.V., Hanover, Lower Saxony

IPD SHARING:
Plan to Share IPD: No